CLINICAL TRIAL: NCT01102920
Title: Health Behaviour Modifications in Obstructive Sleep Apnea. Tailored Behavioural Medicine Strategies to Promote Physical Activity and Weight Loss.
Brief Title: Life-style Changes in Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Research Council (Other Government); Uppsala County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K2008-70X-20838-01-3 PÅ; UU OSA (Other: Uppsala University)
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Sleep Apnea, Obstructive; Obesity
Keywords: Obstructive sleep apnea; Obesity; Behavioural medicine; Physical therapy; Health behaviour change; Physical activity; Eating habits
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity; Motor Activity; Feeding Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored behavioural treatment and CPAP (Experimental): Tailored behavioural treatment targeting physical activity and eating habits.
  Interventions: Behavioral: Behavioural strategies to promote physical activity and weight loss
- CPAP-treatment (Active Comparator): CPAP-treatment as usual. Advice about benefits of physical activity and weight loss.
  Interventions: Device: CPAP

INTERVENTIONS:
Behavioral: Behavioural strategies to promote physical activity and weight loss — 8-10 sessions, 2-4 booster sessions Behavioural protocol in seven steps to initiate, carry out and maintain health-enhancing physical activity and sound eating habits.
  Steps are standardized including: progressive goal setting, self-monitoring, functional behavioural analysis, skills training (basic and applied), generalization, and maintenance and relapse prevention. Content within each step is tailored to individual expectations and skills.
  Treatments are provided by a physical therapist and a dietician.
  Arms: Tailored behavioural treatment and CPAP
Device: CPAP — CPAP-treatment as usual (during nights)
  Arms: CPAP-treatment

SUMMARY:
The primary aim is to study whether a tailored behavioural medicine intervention addressing physical activity and eating habits have additional effects to continuous positive airways pressure (CPAP) in patients with moderate or severe obstructive sleep apnea syndrome (OSAS) combined with obesity. Direct everyday life consequences (see below) of OSAS are studied, as well as cognitive functions and ventilatory parameters. Long-term benefits will be examined in terms of quality of life and everyday life activity. Another aim is to study mechanisms of treatment effects, if any.

The specific goals are:

1. To study changes in OSAS ventilatory parameters following a tailored behavioural medicine intervention addressing physical activity and eating habits (including CPAP) compared to regular CPAP-treatment
2. To study immediate and long-term effects on daytime sleepiness, attention and concentration, everyday life activity, quality of life following a tailored behavioural medicine intervention addressing physical activity and eating habits (including CPAP) compared to regular CPAP-treatment
3. To study associations of changes in metabolic parameters and systemic inflammation and physical activity level and adherence to CPAP-regimen respectively.
4. To identify mediators, moderators, and predictors of treatment effects, if any.

DETAILED DESCRIPTION:
OSAS is characterised by loud snoring, upper airway obstruction, and occasional apnea during sleep. OSAS may affect at least 4% of the men and 2% of the women in middle-age. In Sweden, prevalence figures of 200 000 have been reported. The mechanisms behind OSAS is not fully explained but functionally impaired upper airways muscles, causing a reduction in tonic and phasic contraction during sleep, are proposed one key explanation. The reduced contractions cause partial or complete occlusion of airflow, which in turn cause oxygen desaturation and sleep fragmentation. Patients commonly report everyday life consequences including loud snoring, sleep disturbances, daytime sleepiness, reduced alertness and concentration, and involvement in motor vehicle accidents. Between 7% and 70% of patients suffer from depression and anxiety (figures vary extensively because of methodological differences in existing studies). Due to cardiovascular consequences, OSAS is also linked to hypertension, myocardial infarction, and stroke. Approximately 75% of patients with severe OSAS carry overweight. First line measures recommended for OSAS are conservative including lifestyle modifications, CPAP, and oral appliances. Current state-of-science concludes that CPAP is best possible evidence-based treatment. Despite the use of life style modification recommendations in terms of physical activity and weight loss in accepted guidelines of OSAS, randomised clinical trials supporting these recommendations are rare. Hence, the value of health behaviour modifications has yet to be established. Research within this area is therefore of major interest and urgency, which has motivated the present study design.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe obstructive sleep apnea syndrome (AHI/DI>15)
* BMI>30
* Literate in Swedish language

Exclusion Criteria:

* Physically active patients (walking, bicycling for more than 30 minutes per day,during more than 5 days per week)
* Cardiovascular diseases including myocardial infarctions and stroke
* Patients on waiting list for gastric by-pass

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-05; Primary Completion 2012-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Ventilatory parameters | Baseline, immediate post-treatment, 18-month follow-up
  Ventilatory monitoring at night. Oxygen saturation continuously measured by a pulse oximeter. The following parameters are analysed:
  * desaturation index
  * apnoea-hypnoea index
  * average oxygen saturation during sleep
  * minimum oxigen saturation
  * respiration
  * thoracic respiratory movements
  * snoring
  * heart rate
  * body position

SECONDARY OUTCOMES:
Daytime sleepiness | Baseline, immediate post-treatment, 18-month follow-up
  Epworths sleepiness scale
Attention and concentration | Baseline, immediate post-treatment, 18-month follow-up
  * COWAT
  * Repetition of figures from WAIS
Health-related quality of life | Baseline, immediate post-treatment, 18-month follow-up
  SF-36
Patients' priorities of daily activities and participation | Baseline, immediate post-treatment, 18-month follow-up
  The Patient Goal Priority Questionnaire
Physical activity | Baseline, immediate post-treatment, 18-month follow-up
  * Sensewear armband
  * Physical activity diary
Functional physical capacity | Baseline, immediate post-treatment, 18-month follow-up
  6 minutes walking distance
Eating behaviour | Baseline, immediate post-treatment, 18-month follow-up
  Dutch eating behaviour questionnaire
Self-efficacy and readiness to change behaviour | Baseline, mid-treatment, immediate post-treatment, 18-month follow-up
  * Exercise self-efficacy scale
  * Self-efficacy for sound eating habits
  * Readiness to change behaviour
Anthropometrics | Baseline, immediate post-treatment, 18-month follow-up
  * BMI
  * Waist measurement
  * Neck circumference
Depression | Baseline, immediate post-treatment, 18-month follow-up
  MADRS Depression scale
Fear of movement | Baseline, mid-treatment, immediate post-treatment, 18-month follow-up
  Selected items from the Tampa Scale of Kinesiophobia
Blood sample | Baseline, immediate post-treatment, 18-month follow-up
  * CRP
  * TNF-alfa
  * lgF-1
  * Hb
  * HbA1C
  * s-cholesterol, HDL, LDL, s-triglycerids
  * K, Na
  * Creatinin, Leptin, Sysozym, n-terminal pBNP

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Åsenlöf, Professor, Principal Investigator — Department of Neuroscience, Uppsala University
Locations (1):
- Uppsala University and University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Sporndly-Nees S, Asenlof P, Lindberg E, Emtner M, Igelstrom H. Effects on obstructive sleep apnea severity following a tailored behavioral sleep medicine intervention aimed at increased physical activity and sound eating: an 18-month follow-up of a randomized controlled trial. J Clin Sleep Med. 2020 May 15;16(5):705-713. doi: 10.5664/jcsm.8322. Epub 2020 Feb 6. PMID 32024584